CLINICAL TRIAL: NCT04546477
Title: Prospective, Multicenter, Post-market, Single Arm Study to Confirm the Performance of the RenzanTM Peripheral Stent System in Treating Superficial Femoral and/or Popliteal Artery Disease
Brief Title: Prospective Multicenter Study to Confirm the Performance of the Renzan Stent in Treatment of SFA/POP Artery Disease
Acronym: PRIZER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T134E5
Record Dates: First submitted 2020-02-06; First posted 2020-09-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Superficial Femoral Artery Disease; Popliteal Artery Disease
Keywords: Femoropopliteal; Peripheral intervention; Peripheral stent system

STUDY DESIGN:
Intervention Model Description: Peripheral Stent placement at the location of the initially stenosed or occluded femoropopliteal lesion after proper (1:1 to the reference vessel diameter) vessel preparation without the use of adjunctive debulking devices. Proper vessel preparation should result in ≤20% residual stenosis (as per operator's assessment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): 135 patients stratified into 2 groups:
  * FEM-POP patients: SFA-P1
  * Isolated POP Patients: P1, P2, P3 only
  It is expected the majority of enrolled patients to be FEM-POP category. In case sufficient Isolated POP patients are enrolled, a sub-analysis will be performed on this group of patients.
  Interventions: Device: Stent implantation

INTERVENTIONS:
Device: Stent implantation — Procedure can be conducted via either contralateral or antegrade approach. After a successful target lesion crossing, predilate the lesion using either plain old balloon angioplasty (POBA) or (if necessary) any available specialty balloon. The inflated diameter of the balloon should approximate the diameter of the vessel just distal to the lesion. Proper vessel preparation should achieve diameter of 1:1 to healthy vessel (with ≤20% residual stenosis, as per operator's assessment). Adjunctive debulking devices are prohibited.
  Final stent selection should be confirmed after a proper vessel preparation, considering the reference vessel diameter (RVD) for the optimal 1:1 stent-to-vessel sizing. The implanted dual layer length would encompass the entire lesion with the micromesh, covering it from healthy to healthy tissue. Post-dilatation of the stent for more optimal placement may be done at operator's discretion, using standard angioplasty with uncoated balloon.

SUMMARY:
The primary objective of this study is to confirm the safety and efficacy of the RenzanTM Peripheral Stent System when used for treatment of superficial femoral (SFA) and/or popliteal (POP) artery disease.

This trial plans to include 135 patients in (up to) 10 locations around in Europe.

DETAILED DESCRIPTION:
PRIZER Study is a prospective, multicenter, post-market, single arm study with plan to include approximately 135 patients eligible to be treated with RenzanTM Peripheral Stent System stratified in 2 groups: 90 FEM-POP patients (From superficial femoral Artery to the Proximal edge of patella) and 45 Isolated POP patients (From Hunter's canal to the Origin of anterior tibial artery).

The sponsor will work in accordance with standard operating procedures (SOP) and the Monitoring Plan in order to ensure adherence to the CIP and applicable regulations at the investigational sites.

The Monitoring Plan is built according to a risk-based monitoring approach and describes the level of source data verification to be performed by the monitors.

Risk-based monitoring approach uses all available means to supervise the trial (central monitoring, remote monitoring and on-site monitoring), focusing in critical data points and issues ensuring that adequate monitoring (central, remote and on-site) at each site is completed to ensure protection of the rights and safety of the subjects and the quality and integrity of the data collected and submitted.

The sponsor shall provide training and the necessary guidelines to assist each investigational site on the data collection in the eCRF. Each site is responsible to report the available data requested by the CIP. In order to ensure data quality and avoid missing information in the eCRF, edit checks are designed during database development. In addition, Sponsor's CRA and Data Management team will be responsible to review the data and raise queries accordingly into the eCRF. An audit trail logging all data entered and edited is available within the EDC system. All source documents are maintained in the hospital files ready for inspection by the Sponsor and regulatory authorities upon request. The Sponsor will inform the investigator of the time period for retaining these records as per applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Subject must provide written informed consent prior to the treatment of the target lesion.
3. Subject must be willing to comply with the specified follow-up evaluation schedule.
4. Subject with Rutherford-Becker clinical classification category 2 to 5, with a resting ankle-brachial index (ABI) ≤ 0.9.
5. A superficial femoral and/or popliteal artery lesion with > 50% stenosis or total occlusion.
6. Stenotic or occluded lesion(s) within the same vessel (one long or multiple serial lesions treatable with one stent) ≥ 40 mm and ≤ 140 mm in length, with reference vessel diameter (RVD) ≥ 4.0 mm and ≤ 7.0 mm by visual assessment.
7. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of ipsilateral iliac lesions); Successful ipsilateral iliac artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication, either with PTA or stenting.
8. The target lesion(s) can be successfully crossed with a guide wire and dilated up to 1:1 to healthy vessel (as per operator's assesment).
9. At least one patent native outflow artery (anterior or posterior tibial or peroneal) to the foot, free from significant (≥50%) stenosis (as confirmed by angiography), that has not previously been revascularized. The remaining outflow arteries requiring treatment during the same procedure may be treated only with uncoated devices and before the target lesion.
10. A subject with bilateral obstructive SFA disease is eligible for enrollment into the study. If a subject with bilateral disease is enrolled, the target limb will be selected at the Investigator's discretion, who may use the criteria of lesion length, percent stenosis, and/or calcification content. The contra-lateral procedure should not be done until at least 30 days after the index procedure; however, if contralateral treatment is performed prior to treatment of the target lesion it should be performed at least 1 day before the index procedure with uncoated devices only.
11. The subject is eligible for surgical repair, if necessary.

Exclusion Criteria:

1. Subject has Rutherford-Becker classification category 6.
2. Treatment of lesions requiring the use of adjunctive debulking devices.
3. The use of drug-coated balloons at any step of the procedure.
4. Required stent placement via a popliteal approach.
5. Required stent placement across or within 0.5 cm of the superficial and profunda femoral artery bifurcation.
6. In-stent restenosis treatment or any other procedure which requires stent-in-stent placement to obtain patency.
7. Restenotic lesion that had previously been treated by atherectomy, laser or cryoplasty within 3 months of the index procedure.
8. Lesion with the length that would require stent overlap.
9. Required stent placement within 1 cm of a previously deployed stent.
10. Any significant vessel tortuosity or other parameters prohibiting access to the lesion and/or preventing the stent delivery.
11. Subject with coronary intervention performed less than 90 days prior to or planned within 30 days after the treatment of the target lesion.
12. Known allergies or intolerance to nitinol (nickel titanium), or contrast agent.
13. Any contraindication or known unresponsiveness to dual antiplatelet therapy (DAPT) or anticoagulation therapy.
14. Presence of acute thrombus prior to crossing the lesion.
15. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
16. Thrombophlebitis or deep venous thrombus, within the previous 30 days.
17. Subject receiving dialysis within the previous 30 days.
18. Stroke within the previous 90 days.
19. Known or suspected active infection at the time of the procedure.
20. Subject is pregnant or of child bearing potential
21. Subject has life expectancy of less than 1 year.
22. Subject is participating in an investigational study that has not reached primary endpoint at the time of study screening.
23. Treatment of outflow arteries (anterior or posterior tibial or peroneal) following target lesion treatment (unless bailout).
24. In France: Vulnerable patients, patients deprived from liberty and patients with a physical or mental state altered by disease, age or disability which impacts their ability to defend their interests and for which protection measures are taken ("protected majors" as per French law: articles L1121-5, 6, 8 et L1122-1-3, du code de la santé publique)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-06-24 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint - Death | 30 days
  Freedom from death.
Primary efficacy endpoint - TLR | 30 days
  Freedom from Target Lesion Revascularization (TLR).
Primary efficacy endpoint - Amputation | 30 days
  Freedom from any amputation of the index limb.
Primary efficacy endpoint | 12 months
  Primary patency of the artery at 12 months, defined as no evidence of restenosis or occlusion within the originally treated lesion based on a centrally-read Color Flow Doppler ultrasound in the absence of target lesion revascularization (TLR) (excluding TLR due to thrombosis within 30 days)

SECONDARY OUTCOMES:
Device Success | Intraoperative
  Defined as a successful device deployment according to IFU.
Technical Success | Intraoperative
  Defined as achievement of a final target lesion residual diameter stenosis of <30% based on angiography.
Procedural Success | Intraoperative
  Defined as technical and device success without procedural complication.
Any death | at 1, 6, 12, 24, 36 months
  Cardiovascular death and Non-cardiovascular death
Ankle-brachial Index (ABI) on target limb | at baseline, 1, 6, 12, 24 and 36 months
  Defined as a ratio of the highest ankle systolic blood pressure in one leg, usually measured with a 10 cm cuff at the ankle and using a continuous wave Doppler to detect return of blood flow in the anterior tibial and posterior tibial arteries, to the highest of either arm systolic blood pressure. Performed at rest with subject in supine position.
Clinically-driven Target Lesion Revascularization (CD-TLR) | at 1, 6, 12, 24 and 36 months
  Defined as any TLR associated with deterioration of patient's Rutherford category and/or increase in size of pre-existing ischemic wounds and/or occurrence of new wounds.
Target Lesion Revascularization (TLR) | at 1, 6, 12, 24 and 36 months
  Defined as any repeat percutaneous intervention or bypass surgery performed on the target lesion (including 5mm proximal and distal from the implanted stent).
Target Vessel Revascularization (TVR) | at 1, 6, 12, 24 and 36 months
  Defined as any repeat percutaneous intervention or bypass surgery performed on the target vessel.
Patency of the target lesion | at 6, 24 and 36 months
  Defined as no evidence of restenosis or occlusion within the originally treated lesion based on a centrally-read Color Flow Doppler ultrasound in the absence of target lesion revascularization (TLR) (excluding TLR due to thrombosis within 30 days). Occlusion and restenosis were defined as no color flow or an increase in peak systolic velocity ratio (PSVR) of ≥ 2.4 when compared to the proximal normal segment, respectively.
Limb Ischemia Improvement | at 1, 6, 12, 24 and 36 months
  Defined as an improvement in the Rutherford-Becker Clinical Improvement Scale of greater than or equal to 1.
Major Adverse Events (MAE) | at 1, 6, 12, 24 and 36 months
  Defined as a composite rate of:
  * cardiovascular death
  * procedure-related arterial rupture
  * acute limb ischemia
  * stent thrombosis
  * clinically apparent distal embolization
  * target limb amputation
  * procedure-related bleeding event requiring transfusion
Index Limb Amputations | at 1, 6, 12, 24 and 36 months
  Defined as the surgical removal of tissue anywhere from the toe to hip.
Quality of Life (QoL) | at baseline, 1, 6, 12, 24 and 36 months
  Quality of Life (QoL) assessed as per EQ-5D questionnaire
Walking performance | at baseline, 1, 6, 12, 24 and 36 months
  Walking performance assessed as per Walking Impairment Questionnaire (WIQ)
Rutherford-Becker Scale | at baseline, 1, 6, 12, 24 and 36 months
  Category 0 = Asymptomatic, no hemodynamically significant occlusive disease, Category 1 = Mild claudication, Category 2 = Moderate claudication, Category 3 = Severe claudication, Category 4 = Ischemic rest pain, Category 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, Category 6 = Major tissue loss, extending above trans metatarsal level, functional foot no longer salvageable.
Clinical Improvement | at 1, 6, 12, 24 and 36 months
  Clinical Improvement compared with baseline as per Rutherford-Becker Clinical Improvement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, Dr, Principal Investigator — AZ Sint-Blasius Dendermonde; Torsten Fuss, Dr, Principal Investigator — Elblandhospital Radebeul; Michael Lichtenberg, Dr, Principal Investigator — Karolinen-Hospital: Klinikum Arnsberg; Jérôme Brunet, Dr., Principal Investigator — Clinique Rhône-Durance
Locations (13):
- Belgium (4):
  - AZ Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - Onze Lieve Vrouw (OLV) Ziekenhuis, Aalst
  - Imelda ziekenhuis, Bonheiden
  - Ziekenhuis Oost Limburg, Genk
- France (3):
  - Clinique Rhône-Durance, Avignon
  - Hôpital Paris Saint-Joseph, Paris
  - Clinique Saint Jean - Sud de France, Saint-Jean-de-Védas
- Germany (3):
  - Klinikum Hochsauerland Karolinen-Hospital Hüsten, Arnsberg
  - CCB MVZ Frankfurt und Main-Taunus GbR, Frankfurt
  - Elblandklinikum Radebeul, Radebeul
- Diakonessenhuis, Utrecht, Netherlands
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Cruces, Bilbao

IPD SHARING:
Plan to Share IPD: No